CLINICAL TRIAL: NCT04468308
Title: Assessment of Vision-related Quality of Life (VRQOL) in Cataract Patients During the COVID-19 Pandemic
Brief Title: VRQOL in Cataract Patients During the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: VRQOL Cataract COVID-19
Record Dates: First submitted 2020-06-22; First posted 2020-07-13 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-06

CONDITIONS: Senile Cataract
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Senile Cataract: Patient with senile cataract, whose cataract surgery was postponed in the COVID-19 pandemic
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients complete the National Eye Institute Visual Function Questionnaire 25 pre-operative, 1 month and 3 month postoperatively.

SUMMARY:
The aim of this questionnaire survey is to evaluate the improvement in vision-related quality of life before and after cataract surgery using the National Eye Institute Visual Function Questionnaire 25 and the delay of improvement in the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Senile cataract
* Indication for unilateral or bilateral cataract surgery
* Postponed cataract surgery due to the COVID-19 pandemic
* Signed and dated declaration of consent

Exclusion Criteria:

* Complex form of cataract (traumatic cataract, secondary cataract after intraocular inflammation)
* Amblyopia on the eye that is to be operated on
* Severe, visually impairing eye disease on the eye that is to operated on
* Known dementia or memory problems

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with senile cataract with indication for for unilateral or bilateral cataract surgery.
Sampling Method: Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Improvement Vision-related quality of life | 3 months
  Extent of improvement of vision-related qualitiy of life due to cataract surgery measured with the National Eye Institut Visual Function Questionnaire 25.

SECONDARY OUTCOMES:
Delay of Vision-related quality of life | 3 months
  Delay of improvement of vision-related qualitiy of life in the COVID-19 pandemic measured in days between the originally scheduled operation and the actual operation date
Visual acuity | 1 month
  Visual acuity difference between visual acuity at the time of indication for cataract surgery, on the day of surgery and one month postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No